CLINICAL TRIAL: NCT04394182
Title: Low Doses of Lung Radiation Therapy in Cases of COVID-19 Pneumonia: Prospective Multicentric Study in Radiation Oncology Centers
Brief Title: Ultra Low Doses of Therapy With Radiation Applicated to COVID-19
Acronym: ULTRA-COVID
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Fundacion GenesisCare (Network)
Collaborators: Hospital La Milagrosa (Unknown); Hospital Vithas Valencia Consuelo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20.4.1597-GHM
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pneumonia, Viral; Cytokine Storm
Keywords: Low Dose Radiotherapy; COVID19 pneumonia; Anti-inflammatory effects; Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Pneumonia, Viral; Cytokine Release Syndrome; Respiratory Distress Syndrome | interventions — Oxygen Inhalation Therapy; Lopinavir; lopinavir-ritonavir drug combination; Hydroxychloroquine; Azithromycin; Piperacillin, Tazobactam Drug Combination; Heparin, Low-Molecular-Weight; Adrenal Cortex Hormones; Methylprednisolone; tocilizumab

STUDY DESIGN:
Intervention Model Description: an experimental group will receive ultra low-dose lung radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An experimental group receiving radiotherapy (Experimental): an experimental group with a poor or no response to standard medical treatment and without invasive mechanical ventilation (IMV) will receive ultra low-dose lung radiotherapy (0.8 Gy single dose)
  Interventions: Radiation: Ultra-Low-dose radiotherapy; Device: ventilatory support with oxygen therapy; Drug: Lopinavir/ritonavir; Drug: Hydroxychloroquine; Drug: Azithromycin; Drug: Piperacillin/tazobactam; Drug: Low molecular weight heparin; Drug: Corticosteroid injection; Drug: Tocilizumab

INTERVENTIONS:
Radiation: Ultra-Low-dose radiotherapy — The total dose to be administered was 0.8 Gy in an only single session including both whole-lungs extended 1cm isometric in all directions.
Device: ventilatory support with oxygen therapy — Oxygen Therapy: Nasal Cannula (NC); Ventimask (VMK) or VMK with reservoir
Drug: Lopinavir/ritonavir — 100/400 mg/12h; 7-10 days
  Other Names: Kaletra
Drug: Hydroxychloroquine — 200 mg/12h
  Other Names: Dolquine
Drug: Azithromycin — 500 mg/24h, 3 days
Drug: Piperacillin/tazobactam — 4 g / 0.5 g administered every 6-8 hours through a vein (directly into the bloodstream), for 5-14 days. Adjustment to kidney function
Drug: Low molecular weight heparin — prophylactic doses
Drug: Corticosteroid injection — 250mg x 3 boluses
  Other Names: Urbason
Drug: Tocilizumab — 600mg single dose

SUMMARY:
The host response against the coronavirus 2 (SARS-CoV-2) appears to be mediated by a 'cytoquine storm' developing a systemic inflammatory mechanism and an acute respiratory distress syndrome (ARDS), in the form of a bilateral pneumonitis, requiring invasive mechanical ventilation (IMV) in an important group of patients.

In terms of preventing progression to the critical phase with the consequent need of admission to the intensive care units (ICU), it has been recently proposed that this inflammatory cytoquine-mediated process can be safely treated by a single course of ultra-low radiotherapy (RT) dose < 1 Gy.

The main purpose of the study was to analyze the efficacy of ultra low-dose pulmonary RT, as an anti-inflammatory intention in patients with SARS-Cov-2 pneumonia with a poor or no response to standard medical treatment and without IMV.

DETAILED DESCRIPTION:
The exceedingly high mortality rates of severe and critical COVID-19 warrant the evaluation of novel therapies that could potentially mitigate the advanced disease manifestations. In this context, is proposes a prospective multicenter study. It will include 15 patients, to assess the feasibility and efficacy of low-dose lung irradiation in COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years-old.
2. Diagnosis of pneumonia due to COVID-19 serologically proven by polymerase chain reaction (PCR) or highly suspected to be COVID-related.
3. Charlson Comorbidity Index (CCI) less than 6 score.
4. Poor or no response to standard medical treatment, based on:

   *% Sat02 <93%
   * Oxygen therapy escalation (Understanding from less to more need for support: Nasal Cannula-NC-; Ventimask -VMK- and VMK with reservoir)
   * Pa02 / Fi02 (blood gas analysis) <300 mmHg
   * 1 or more inflammatory and immunological analytical parameters such as lymphocytes, IL-6, D-dimer, ferritin, LDH, C Reactive Protein (CRP) and fibrinogen with values above the normal range, except lymphocytes.
   * Radiological impairment defined as worsening of TSS throughout admission or score at admission: TSS> 5 by a diagnostic baseline CT scan.
5. Eastern Cooperative Oncology Group (ECOG) Status < or = 3
6. Life expectancy (LE)> 1 month at hospital admission for COVID-19
7. No previous thoracic RT (relative-individualization criteria) or chemotherapy (chemoinduced pulmonary toxicity, eg Bleomycin).
8. Verbal information on the procedure, objective and secondary effects, acceptance and signing of informed consent by the patient or legal guardian.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* Any uncontrolled intercurrent illness that would put the patient at greater risk or limit compliance with study requirements in the opinion of the investigator.
* Patients admitted in ICU.
* Refusal of treatment after verbal information.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-03-21 (Estimated)

PRIMARY OUTCOMES:
Oxygen Therapy Status at Day 2 | At 2 after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through clinical evaluation.It was performed by oxygen therapy status assessment after RT treatment. Improvement criteria is considered as an oxygen therapy de-escalation (more to less need for support: Ventimask (VMK) with reservoir >VMK >Nasal Cannula-(NC).)
Oxygen Saturation (Sat02; Pulse oximeter measurement) at Day 2 | At 2 days after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through clinical evaluation. .It was performed by oxygen saturation (Sat02 %) status assessment after RT treatment. Improvement criteria is considered as a Sat02 with/without oxygen therapy >93% (Pulse oximeter measurement)

SECONDARY OUTCOMES:
Blood Gas Analysis at Day 2 | At 2 days after RT
  Pa02 / Fi02 > 300 mmHg
Blood Test at Day 2 | At 2 days after RT
  Achievement of normal range value in 1 or more of the inflammatory and immunological parameters (lymphocytes, IL-6, D-dimer, ferritin, LDH, C Reactive Protein (CRP) and fibrinogen)
Oxygen Therapy Status at Day 5 | At 5 after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through clinical evaluation.It was performed by oxygen therapy status assessment after RT treatment. Improvement criteria is considered as an oxygen therapy de-escalation (more to less need for support: Ventimask (VMK) with reservoir >VMK >Nasal Cannula-(NC).)
Oxygen Saturation (Sat02; Pulse oximeter measurement) at Day 5 | At 5 days after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through clinical evaluation. .It was performed by oxygen saturation (Sat02 %) status assessment after RT treatment. Improvement criteria is considered as a Sat02 with/without oxygen therapy >93% (Pulse oximeter measurement)
Blood Test at Day 5 | At 5 days after RT
  Achievement of normal range value in 1 or more of the inflammatory and immunological parameters (lymphocytes, IL-6, D-dimer, ferritin, LDH, C Reactive Protein (CRP) and fibrinogen)
Oxygen Therapy Status at Day 7 | At 7 after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through clinical evaluation.It was performed by oxygen therapy status assessment after RT treatment. Improvement criteria is considered as an oxygen therapy de-escalation (more to less need for support: Ventimask (VMK) with reservoir >VMK >Nasal Cannula-(NC).)
Oxygen Saturation (Sat02; Pulse oximeter measurement) at Day 7 | At 7 days after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through clinical evaluation. .It was performed by oxygen saturation (Sat02 %) status assessment after RT treatment. Improvement criteria is considered as a Sat02 with/without oxygen therapy >93% (Pulse oximeter measurement)
Blood Test at Day 7 | At 7 days after RT
  Achievement of normal range value in 1 or more of the inflammatory and immunological parameters (lymphocytes, IL-6, D-dimer, ferritin, LDH, C Reactive Protein (CRP) and fibrinogen)
Change from baseline Total Severity Score (TSS) analyzed in a thoracic CT scan at Day 7 | At 7 days after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through radiological evaluation.It was performed by thoracic CT scan after RT treatment .
  It is considered a radiological improvement the decrease of the Total Severity Score (TSS) from the baseline in > or = 1 point.
  NOTE: The score values ranged from 0 to 4 according to the sum of the percentage involvement of each of the 5 lung lobes. The total severity score (TSS), was reached by summing the overall involvement in the lung (0-20 points)
Recovery time | From RT administration until hospital discharge or death
  Recovery time after RT administration until hospital discharge or death (<48h; 2-7 days; >7 days; clinical worsening or death)
COVID-19 status | At 7 days after RT
  COVID-19 negativization test
Change from baseline Total Severity Score (TSS) analyzed in a thoracic CT scan al Month 1 | At 1 month after RT
  To evaluate the efficacy of ultra low-dose pulmonary RT through radiological evaluation.It was performed by thoracic CT scan after RT treatment .
  It is considered a radiological improvement the decrease of the Total Severity Score (TSS) from the baseline in > or = 1 point.
  NOTE: The score values ranged from 0 to 4 according to the sum of the percentage involvement of each of the 5 lung lobes. The total severity score (TSS), was reached by summing the overall involvement in the lung (0-20 points)
Acute Toxicity | 1-3 months after RT
  Toxicity was assessed and rated according to the NIH Common Terminology Criteria for Adverse Events (CTCAE version 5.0) and RTOG scales.

CONTACTS AND LOCATIONS:
Overall Officials: Escarlata López Ramírez, MD, PhD, Principal Investigator — Fundacion GenesisCare
Locations (2):
- Spain (2):
  - Hospital La Milagrosa, GenesisCare, Madrid
  - Hospital Vithas Valencia Consuelo, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Medical history and biographical and clinical data of each patient will be recorded and shared.
  The overall results of any research conducted will be available on study data publication.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Result] Kirkby C, Mackenzie M. Is low dose radiation therapy a potential treatment for COVID-19 pneumonia? Radiother Oncol. 2020 Jun;147:221. doi: 10.1016/j.radonc.2020.04.004. Epub 2020 Apr 6. No abstract available. PMID 32342871
- [Result] Berk LB, Hodes PJ. Roentgen therapy for infections: an historical review. Yale J Biol Med. 1991 Mar-Apr;64(2):155-65. PMID 1750226
- [Result] Calabrese EJ, Dhawan G. How radiotherapy was historically used to treat pneumonia: could it be useful today? Yale J Biol Med. 2013 Dec 13;86(4):555-70. PMID 24348219
- [Result] Cuttler JM. Application of Low Doses of Ionizing Radiation in Medical Therapies. Dose Response. 2020 Jan 6;18(1):1559325819895739. doi: 10.1177/1559325819895739. eCollection 2020 Jan-Mar. PMID 31933547
- [Result] Arenas M, Sabater S, Hernandez V, Rovirosa A, Lara PC, Biete A, Panes J. Anti-inflammatory effects of low-dose radiotherapy. Indications, dose, and radiobiological mechanisms involved. Strahlenther Onkol. 2012 Nov;188(11):975-81. doi: 10.1007/s00066-012-0170-8. Epub 2012 Aug 22. PMID 22907572
- [Result] Calabrese EJ, Dhawan G, Kapoor R, Kozumbo WJ. Radiotherapy treatment of human inflammatory diseases and conditions: Optimal dose. Hum Exp Toxicol. 2019 Aug;38(8):888-898. doi: 10.1177/0960327119846925. Epub 2019 May 6. PMID 31060383
- [Result] Rodel F, Keilholz L, Herrmann M, Sauer R, Hildebrandt G. Radiobiological mechanisms in inflammatory diseases of low-dose radiation therapy. Int J Radiat Biol. 2007 Jun;83(6):357-66. doi: 10.1080/09553000701317358. PMID 17487675
- [Result] Schaue D, Jahns J, Hildebrandt G, Trott KR. Radiation treatment of acute inflammation in mice. Int J Radiat Biol. 2005 Sep;81(9):657-67. doi: 10.1080/09553000500385556. PMID 16368644
- [Result] Torres Royo L, Antelo Redondo G, Arquez Pianetta M, Arenas Prat M. Low-Dose radiation therapy for benign pathologies. Rep Pract Oncol Radiother. 2020 Mar-Apr;25(2):250-254. doi: 10.1016/j.rpor.2020.02.004. Epub 2020 Feb 22. PMID 32140081
- [Result] Lara PC, Burgos J, Macias D. Low dose lung radiotherapy for COVID-19 pneumonia. The rationale for a cost-effective anti-inflammatory treatment. Clin Transl Radiat Oncol. 2020 Apr 25;23:27-29. doi: 10.1016/j.ctro.2020.04.006. eCollection 2020 Jul. PMID 32373721
- [Derived] Moreno-Olmedo E, Suarez-Gironzini V, Perez M, Filigheddu T, Minguez C, Sanjuan-Sanjuan A, Gonzalez JA, Rivas D, Gorospe L, Larrea L, Lopez E. COVID-19 pneumonia treated with ultra-low doses of radiotherapy (ULTRA-COVID study): a single institution report of two cases. Strahlenther Onkol. 2021 May;197(5):429-437. doi: 10.1007/s00066-020-01743-4. Epub 2021 Jan 27. PMID 33502567
- See also: Li, K., Fang, Y., Li, W. et al. CT image visual quantitative evaluation and clinical classification of coronavirus disease (COVID-19). Eur Radiol (2020). https://doi.org/10.1007/s00330-020-06817-6 — https://doi.org/10.1007/s00330-020-06817-6